CLINICAL TRIAL: NCT02260154
Title: Effectiveness of Duspatalin® (Mebeverine Hydrochloride) 200 mg b.i.d. in Patients With Post-cholecystectomy Gastrointestinal Spasm: a Post Marketing Observational Program in the Russian Federation
Brief Title: Effectiveness of Duspatalin® in Patients With Post-cholecystectomy Gastrointestinal Spasm
Acronym: ODYSSEY
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: MEBE5002
Record Dates: First submitted 2014-09-29; First posted 2014-10-09 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-03

CONDITIONS: Post-cholecystectomy Gastrointestinal Spasms
Keywords: Duspatalin; mebeverine; cholecystectomy; gastrointestinal spasm; abdominal pain; dyspepsia; antispasmodics
MeSH Terms: conditions — Abdominal Pain; Dyspepsia | interventions — mebeverine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post-cholecystectomy gastrointestinal spasms: Adult subjects suffering from post-cholecystectomy gastrointestinal spasms not requiring surgical treatment prescribed Duspatalin® 200 mg twice a day
  Interventions: Drug: Mebeverine

INTERVENTIONS:
Drug: Mebeverine — Subjects treated by Duspatalin (mebeverine) 200 mg BID (bis in die = twice a day) upto 6 weeks in accordance with routine practice will be observed
  Other Names: Duspatalin

SUMMARY:
Prospective, multicenter, non-comparative, observational program designed to assess the effectiveness of a 2-6 weeks treatment with Duspatalin® 200mg bis in die = twice a day (BID) and changes in quality of life in patients with post-cholecystectomy gastro-intestinal spasms

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years to 65 years;
* Patients suffering from post-cholecystectomy GI-spasms in the last 3 months with symptom onset at least 6 months prior to inclusion and not requiring surgical treatment;
* Laparoscopic cholecystectomy between 6 months to 5 years before enrollment;
* Patients having been prescribed Duspatalin® (mebeverine) 200 mg BID (bis in die = twice a day) in accordance with approved local label;
* Patient's written authorization to provide data for the program

Exclusion Criteria:

* General and specific contraindications to Duspatalin® treatment according to the local label;
* Planned Endoscopic Retrograde Cholangiopancreatography (ERCP) and/or surgical treatment;
* Being currently treated or having been treated with Duspatalin® within the 6 weeks prior to entering the program;
* Pregnancy or lactation;
* Other conditions that make patient participation impossible (by investigator judgment);
* Previous enrollment in the present program;
* Treatment with other antispasmodics, pain-medication (Nonsteroidal anti-inflammatory drugs (NSAIDs), tramadol, etc.) within 2 weeks prior to inclusion into the observational study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Vladimirova, MD, PhD, Study Director — Abbott
Locations (21):
- Russia (21):
  - Research Facility ID ORG-001035, Chita
  - State Budget Institution " Irkutsk State Medical Academy of postgraduate education", Irkutsk
  - Research Facility ID ORG-001038, Izhevsk
  - Research Facility ID ORG-001033, Kazan'
  - Non-governmental Healthcare Institution "Road Clinical Hospital on the station Khabarovsk-1 OSS "Russian Railways", Khabarovsk
  - Research Facility ID ORG-001034, Krasnoyarsk
  - Research facility ID ORG-001039, Moscow
  - Federal State Budget Institution "Outpatient hospital №1" Administration of the President of the Russian Federation, Moscow
  - State Budget Institution "Pirogov Russian National Research Medical University", on the base of State Budget Institution of Health Care of Moscow "City Clinical Hospital №31", Moscow
  - State Budget Institution "Russian Medical Academy of Postgraduate Studies, Moscow
  - State Budget Institution of Health Care of Moscow region " MF Vladimirsky Moscow Region Scientific Research Clinical University", Moscow
  - Research Facility ID ORG-001024, Moscow
  - State Budget Institution "Nizhny Novgorod Regional Clinical Hospital n.a. Semashko", Nizhny Novgorod
  - State Budget Institution "Novosibirsk State Medical University", Novosibirsk
  - Research Facility ID ORG-000903, Omsk
  - Federal State Budget Institution Hospital of the Pushchino Scientific Center of the Russian Academy of Sciences, Pushchino
  - Research Facility ID ORG-001036, Rostov-on-Don
  - Federal State Budget Institution All-Russian Center of Emergency and Radiation Medicine of EMERCOM of Russia, Saint Petersburg
  - State Budget Institution "North-Western State Medical University named after I.I. Mechnikov", on the base of State Budget Institution "Sity Clinical Hospital #26", Saint Petersburg
  - Research Facility ID ORG-001037, Saransk
  - City Clinical Hospital #40, Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Groups:
- Post-cholecystectomy Gastrointestinal Spasms: Adult subjects suffering from post-cholecystectomy gastrointestinal spasms not requiring surgical treatment prescribed Duspatalin® 200 mg twice a day
  Mebeverine: Subjects treated by Duspatalin (mebeverine) 200 mg bis in die = twice a day (BID) upto 6 weeks in accordance with routine practice will be observed
Period: Overall Study
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Started | 220
Completed | 218
Not Completed | 2
Not completed — Screening failure | 2

BASELINE CHARACTERISTICS:
Population: Adult subjects suffering from post-cholecystectomy gastrointestinal spasms not requiring surgical treatment prescribed Duspatalin® 200 mg twice a day
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 218
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 216
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Russia | 218
Working status [Count of Participants; unit: Participants]
  employed | 137
  unemployed | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage of "Responders" to Duspatalin® Therapy
Description: Patients indicating being 'symptom-free' or 'markedly improved'on Global Patient Assessment
Time Frame: 2 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 218
percentage of participants
  Symptom-free or markedly improved | 63.6 [56.8 to 70.0]
  Other values (slightly improved, unchanged, worse) | 36.4 [30.0 to 43.2]

2. Secondary Outcome: Percentage of "Responders" to Duspatalin® Therapy
Time Frame: Up to 6 weeks
Population: Extended set includes those patients who completed at least 6 weeks treatment of Duspatalin
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 101
percentage of participants | 79.0 [69.7 to 86.5]

3. Secondary Outcome: Changes in Abdominal Pain
Description: Measured by 11-items Numerous Rating Scale where 0 represents no pain and 10 represents the worst pain. Negative change corresponds to better result. Changes are calculated as Week 2 value minus Baseline value and Week 6 value minus Baseline value.
Time Frame: Baseline, 2 weeks and up to 6 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 217
units on a scale
  change from baseline at Week 2 | -3.7 (2.28)
  change from baseline at Week 6 | -4.4 (2.36)

4. Secondary Outcome: Changes in Dyspepsia Symptoms
Description: Measured by 11-items Numerous Rating Scale where 0 represents no symptoms and 10 represents the worst symptoms. Negative change corresponds to better result. Changes are calculated as Week 2 value minus Baseline value and Week 6 value minus Baseline value.
Time Frame: Baseline, 2 weeks and up to 6 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 217
units on a scale
  change from baseline at Week 2 | -2.0 (2.29)
  change from baseline at Week 6 | -2.3 (2.41)

5. Secondary Outcome: Changes in Stool Habits and Percentage of Patients Reporting Abnormal Stool Form
Description: Changes in Stool Habits: The change is presented as the proportion of patients whose Changes in Stool Habits from 'Abnormal' to 'Normal' and vice versa were registered. "Positive" is defined as Change from 'Abnormal stool form at BL' to 'Normal stool form at Week 2'. "Negative" is defined as Change from 'Normal stool form at BL' to 'Abnormal stool form at Week 2'.
Time Frame: Baseline to Week 2
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 217
percentage of participants
  Positive | 38.25
  Negative | 2.30

6. Secondary Outcome: Changes in Quality of Life
Description: Gastrointestinal Quality of Life Index contains 36 questions with 4 possible answers per each (most desirable option returns 4 points, and least desirable option returns 0 points). Total score of the GIQLI is calculated as sum of all items. The source scores are transformed and scaled from 0 to 100. The high score corresponds to better result. Changes are calculated as Week 2 value minus Baseline value and Week 6 value minus Baseline value.
Time Frame: Baseline, 2 weeks and up to 6 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 217
units on a scale
  change from baseline at Week 2 | 16.802 (11.8489)
  change from baseline at Week 6 | 21.737 (13.4339)

7. Secondary Outcome: Health Economic Data
Description: Relevant concomitant medication
Time Frame: Baseline, up to 6 weeks
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 218
percentage of participants
  ACE inhibitors | 9.6
  Alpha adrenoreceptor antagonist | 0.5
  Aluminium compounds | 2.3
  Angiotensine II antagonist | 1.4
  Anti arrhythmics | 0.5
  Anti diarrheal | 1.4
  Anti inflammatory | 0.5
  Barbiturates | 0.5
  Beta blocking against agents, selective | 4.1
  Biguaniges | 0.9
  Bile acid preparations | 10.1
  Bioflavonoids | 0.5
  Blood transfusion, auxilary products | 0.5
  Beta blocking agents, and other antihypertensives | 0.5
  Beta blocking agents, thiazides | 0.5

8. Secondary Outcome: Reasons for Continuing Treatment Beyond 2 Weeks
Description: List and rate of reasons
Time Frame: 2 weeks
Population: Extended Set includes those patients who completed at least 6 weeks treatment of Duspatalin
Measure: Number; unit: percentage of participants
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 101
percentage of participants
  Expectation in higher effectiveness | 84.2
  Tend to treat beyond 2 weeks | 4.0
  Maintenance of achieved effect | 11.9

9. Secondary Outcome: Healths Economic Data 2
Description: Number of visits to clinic for currently employed subjects. Change is calculated as Week 6 value minus Baseline value. Negative change means less number of visits to clinic.
Time Frame: from baseline at Week 6
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 101
number of visits | -0.9 (1.19)

10. Secondary Outcome: Health Economics Data 3
Description: Number of days missed from work for currently employed subjects. Change is calculated as Week 6 value minus Baseline value. Negative change means less number of days missed from work.
Time Frame: change from baseline at Week 6
Population: Adult subjects suffering from post-cholecystectomy gastrointestinal spasms not requiring surgical treatment prescribed Duspatalin® 200mg twice a day
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 57
Number of days | -2.1 (3.48)

11. Secondary Outcome: Changes in Stool Habits and Percentage of Patients Reporting Abnormal Stool Form 2
Description: Changes in Stool Habits: The change is presented as the proportion of patients whose Changes in Stool Habits from 'Abnormal' to 'Normal' and vice versa were registered. "Positive" is defined as Change from 'Abnormal stool form at BL' to 'Normal stool form at Week 6'. "Negative" is defined as Change from 'Normal stool form at BL' to 'Abnormal stool form at Week 6'.
Time Frame: Baseline to Week 6
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Number analyzed (Participants) | 100
percentage of participants
  Positive | 40.00
  Negative | 2.00

ADVERSE EVENTS:
Arm/Group | Post-cholecystectomy Gastrointestinal Spasms
Serious Adverse Events (participants affected / at risk) | 0/218
Other Adverse Events (participants affected / at risk) | 1/218
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post-cholecystectomy Gastrointestinal Spasms (N=218)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less